CLINICAL TRIAL: NCT03761459
Title: Current Surgical Practices and Surgical Site Infection at Ayder Comprehensive Specialized Hospital in Mekelle, Ethiopia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Mekelle University (Other)
Responsible Party: Principal Investigator, Erin Cavanaugh, Assistant Professor, Obstetrics and Gynecology, University of Illinois at Chicago
Other Study IDs: 2017-1251
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Surgical Wound Infection; Infected Wound; Surgical Site Infection; Surgery--Complications; Surgery; Surgical Wound
Keywords: Surgical site infection; low and middle income country; low resource setting; Africa; Ethiopia
MeSH Terms: conditions — Surgical Wound Infection; Wound Infection; Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the current surgical practices at Ayder Comprehensive Specialized Hospital in comparison to the World Health Organization's Surgical Unit Based Safety Programme guidelines and aims to determine how deviations from those guidelines are associated with varying rates of surgical site infection incidence in this population. The results of this study will help elucidate risk factors for surgical site infection and prioritize future interventions to decrease the rate of surgical site infection at Ayder Comprehensive Specialized Hospital, as well as other low and middle-income hospitals. The data collected regarding surgical site infection rates will also prove beneficial in measuring outcomes of any interventions that are developed as a result of this study.

DETAILED DESCRIPTION:
Surgical site infection continues to be a major cause of morbidity and mortality around the world with low and middle-income countries disproportionately affected with rates as high as 30-40% compared to an average rate of less than 3% in high income countries. In addition to the grave clinical implications of these infections, the additional costs incurred by both patients and treating institutions can be catastrophic.

The World Health Organization's "Clean Care is Safer Care" initiated quality improvement projects in five African hospitals between 2013 and 2015, demonstrating that low-cost interventions can decrease the rates of surgical site infection in low and middle-income countries. This successful initiative formed the basis of the World Health Organization's Surgical Unit Based Safety Programme guidelines.

This will be a prospective cohort study collecting data about surgical practices, pre- and post-operative care and post-operative infection from time of admission through post-operative day 30. Patients will be identified when they are scheduled for surgery and undergo consent process. If they consent to participate in the study their clinical course will be followed through post-operative day 30. Inpatient observational data will be collected to determine whether current practices are in line with World Health Organization's Surgical Unit Based Safety Programme guidelines. Potential confounding risk factors for infection will be identified, and post-operative information will be collected through inpatient follow up as well as telephone calls on post-operative day ten and 30 to assess for signs or symptoms of surgical site infection.

ELIGIBILITY:
Inclusion Criteria:

* All patients (male and female) 18 years of age or older undergoing any surgery (elective, scheduled, urgent or emergent) including obstetrics and gynecology cases at ACSH in Mekelle Ethiopia.

Exclusion Criteria:

* Patients under the age of 18.
* Patients who undergo surgery involving permanent implants (as these patients would require follow up for 1 year to effectively rule out surgical site infection and this is beyond the data collection time frame of this study)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Male and female patients 18 years of age or older undergoing any surgical procedure in the main operating theaters at Ayder Comprehensive Specialized Hospital in Mekelle, Ethiopia during the 12-month study period, not including cases involving permanent implants. Inpatient collection of data will occur prospectively with supplemental information recorded from medical records if patient consents. Post-discharge data will be collected for patients who consent for follow-up.
Sampling Method: Probability Sample
Enrollment: 1240 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to World Health Organization (WHO) Surgical Unit based Safety Programme (SUSP) guidelines | 12 months
  Determine whether current surgical practices at Ayder Comprehensive Specialized Hospital (ACSH) follow each of the six components of the WHO SUSP guidelines through prospective data collection via case report form, which is filled out by trained data collector during procedure and during the post-operative period to document whether each of the SUSP guidelines are being followed

SECONDARY OUTCOMES:
Surgical site infection incidence at ACSH | 30 days from operation
  Determine the current surgical site infection rate at ACSH through prospective data collection of operations occurring at ACSH during the study period
Trends between adherence to WHO SUSP guidelines and infection | 12 months
  Evaluate trends between surgical site infection and the adherence to each of the WHO SUSP guideline components using logistic regression analysis of prospectively collected data regarding adherence to WHO SUSP guidelines and occurrence of post-operative infection

CONTACTS AND LOCATIONS:
Overall Officials: Erin Cavanaugh, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Ayder Comprehensive Referral Hospital, Mek'ele, Tigray, Ethiopia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to anyone outside of our study.

REFERENCES:
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Background] Astagneau P, Rioux C, Golliot F, Brucker G; INCISO Network Study Group. Morbidity and mortality associated with surgical site infections: results from the 1997-1999 INCISO surveillance. J Hosp Infect. 2001 Aug;48(4):267-74. doi: 10.1053/jhin.2001.1003. PMID 11461127
- [Background] Kirkland KB, Briggs JP, Trivette SL, Wilkinson WE, Sexton DJ. The impact of surgical-site infections in the 1990s: attributable mortality, excess length of hospitalization, and extra costs. Infect Control Hosp Epidemiol. 1999 Nov;20(11):725-30. doi: 10.1086/501572. PMID 10580621
- [Background] Coello R, Charlett A, Wilson J, Ward V, Pearson A, Borriello P. Adverse impact of surgical site infections in English hospitals. J Hosp Infect. 2005 Jun;60(2):93-103. doi: 10.1016/j.jhin.2004.10.019. PMID 15866006
- [Background] Gaynes RP, Culver DH, Horan TC, Edwards JR, Richards C, Tolson JS. Surgical site infection (SSI) rates in the United States, 1992-1998: the National Nosocomial Infections Surveillance System basic SSI risk index. Clin Infect Dis. 2001 Sep 1;33 Suppl 2:S69-77. doi: 10.1086/321860. PMID 11486302
- [Background] Ngaroua, Ngah JE, Benet T, Djibrilla Y. [Incidence of surgical site infections in sub-Saharan Africa: systematic review and meta-analysis]. Pan Afr Med J. 2016 Jun 29;24:171. doi: 10.11604/pamj.2016.24.171.9754. eCollection 2016. French. PMID 27795768
- [Background] Chu K, Maine R, Trelles M. Cesarean section surgical site infections in sub-Saharan Africa: a multi-country study from Medecins Sans Frontieres. World J Surg. 2015 Feb;39(2):350-5. doi: 10.1007/s00268-014-2840-4. PMID 25358418
- [Background] Amenu D, Belachew T, Araya F. Surgical site infection rate and risk factors among obstetric cases of jimma university specialized hospital, southwest ethiopia. Ethiop J Health Sci. 2011 Jul;21(2):91-100. doi: 10.4314/ejhs.v21i2.69049. PMID 22434989
- [Background] Mengesha RE, Kasa BG, Saravanan M, Berhe DF, Wasihun AG. Aerobic bacteria in post surgical wound infections and pattern of their antimicrobial susceptibility in Ayder Teaching and Referral Hospital, Mekelle, Ethiopia. BMC Res Notes. 2014 Aug 27;7:575. doi: 10.1186/1756-0500-7-575. PMID 25164127
- [Background] Wasihun AG, Zemene Y. Bacterial profile and antimicrobial susceptibility patterns of otitis media in Ayder Teaching and Referral Hospital, Mekelle University, Northern Ethiopia. Springerplus. 2015 Nov 14;4:701. doi: 10.1186/s40064-015-1471-z. eCollection 2015. PMID 26609503
- [Background] Aiken AM, Karuri DM, Wanyoro AK, Macleod J. Interventional studies for preventing surgical site infections in sub-Saharan Africa - A systematic review. Int J Surg. 2012;10(5):242-9. doi: 10.1016/j.ijsu.2012.04.004. Epub 2012 Apr 14. PMID 22510442
- [Background] Teshager FA, Engeda EH, Worku WZ. Knowledge, Practice, and Associated Factors towards Prevention of Surgical Site Infection among Nurses Working in Amhara Regional State Referral Hospitals, Northwest Ethiopia. Surg Res Pract. 2015;2015:736175. doi: 10.1155/2015/736175. Epub 2015 Dec 15. PMID 26788549
- [Background] Aiken AM, Wanyoro AK, Mwangi J, Mulingwa P, Wanjohi J, Njoroge J, Juma F, Mugoya IK, Scott JA, Hall AJ. Evaluation of surveillance for surgical site infections in Thika Hospital, Kenya. J Hosp Infect. 2013 Feb;83(2):140-5. doi: 10.1016/j.jhin.2012.11.003. Epub 2013 Jan 18. PMID 23332563
- [Background] Nguhuni B, De Nardo P, Gentilotti E, Chaula Z, Damian C, Mencarini P, Nicastri E, Fulment A, Piscini A, Vairo F, Aiken AM, Ippolito G. Reliability and validity of using telephone calls for post-discharge surveillance of surgical site infection following caesarean section at a tertiary hospital in Tanzania. Antimicrob Resist Infect Control. 2017 May 8;6:43. doi: 10.1186/s13756-017-0205-0. eCollection 2017. PMID 28503302
- [Background] Hurwitz EE, Simon M, Vinta SR, Zehm CF, Shabot SM, Minhajuddin A, Abouleish AE. Adding Examples to the ASA-Physical Status Classification Improves Correct Assignment to Patients. Anesthesiology. 2017 Apr;126(4):614-622. doi: 10.1097/ALN.0000000000001541. PMID 28212203
- See also: Surveillance of surgical site infections in Europe, 2008-2009 by the European Centre for Disease Prevention and Control — https://ecdc.europa.eu/sites/portal/files/media/en/publications/Publications/120215_SUR_SSI_2008-2009.pdf
- See also: Microbial contamination of operating theatre at Ayder Referral Hospital, Northern Ethiopia. International Journal of Pharma Sciences and Research, 6(10), 1264-1267 — http://www.ijpsr.info/docs/IJPSR15-06-10-013.pdf
- See also: SUSP project in African Surgical Departments — https://www.who.int/news-room/feature-stories/detail/the-surgical-unit-based-safety-programme-(susp)-in-african-hospitals